CLINICAL TRIAL: NCT02049307
Title: Losartan to Reduce Inflammation and Fibrosis Endpoints in HIV Trial
Acronym: LIFE-HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Jason Baker, Protocol Chair, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCC-007
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Inflammation; Fibrosis
MeSH Terms: conditions — Inflammation; Fibrosis | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Losartan 100mg daily
  Interventions: Drug: Losartan 100mg daily
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Losartan 100mg daily
  Arms: Treatment
Drug: Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential effectiveness of losartan (100mg daily) for reducing inflammation and improving immune recovery.

DETAILED DESCRIPTION:
Our general goal is to evaluate the potential effectiveness of losartan (100mg daily) for reducing inflammation and improving immune recovery, given the potential for these treatment effects to reduce risk for long-term non-AIDS-defining complications among older HIV positive participants. Prior to conducting a clinical outcome trial, candidate treatments must be studied among HIV positive patients given the unique pathogenesis driving inflammation and disease risk.

The potential benefits of losartan (100mg daily) will be studied among HIV positive individuals over age 50 years whose CD4 counts remain ≤600 cells/mm3. Participants (n=110, 55 per group) will be randomized to receive losartan or matching placebo daily. After randomization, participants will start losartan (or placebo) at a dose of 50mg once daily, increasing to 100mg once daily at the 2-week study visit pending results of a week 2 toxicity lab evaluation (see 2.4 below for criteria). Following month 1, participants will return for follow-up study visit procedures at months 3, 6, 9, and 12.

Changes from baseline in measures of inflammation, immune activation, immune recovery and fibrosis within lymphatic tissues will be studied. The primary outcome will be the average of IL-6 levels over 12 months, and the main secondary outcome will be change in CD4 count in blood over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection (verified by previous positive antibody or detectable HIV RNA level)
* Age > 50 years
* Receiving continuous ART for >= 2 years (regimen changes > 6 months prior to enrollment are allowed)
* HIV RNA level < 200 copies/mL for >= 1 year (1 measure >= 200 allowed if also < 1000 and preceded and followed by values < 200 copies/mL)
* Blood CD4+ T-cell count < 600 cells/mm cubed
* Systolic blood pressure > 120 mmHg (mean value if >= 2 measures obtained)
* Estimated glomerular filtration rate (GFR )> 30 mL/min/1.73 m squared
* Do not anticipate starting or stopping statin or aspirin therapy during the study

Exclusion Criteria:

* Pregnancy or breastfeeding
* A contra-indication to taking an angiotensin receptor blocker (ARB) (e.g., cirrhosis, prior angioedema with angiotensin-converting enzyme inhibitor (ACE-I), or use of drug with potential drug-interaction [e.g., rifaximin])
* A clinical indication for ARB or ACE-I therapy (e.g., cardiovascular disease (CVD), stroke, or diabetes mellitus (DM))
* Current treatment with ARB or medication with overlapping mechanism (e.g., ACE-I or aldosterone antagonist)
* Current treatment with immunomodulatory drugs within the past 6 months
* Current hepatitis treatments (e.g., interferon, ribavirin) within the past 6 months
* Serum potassium > 5.0 millimoles per liter (mmol/L) within 3 months of entry
* Invasive cancer in the prior year or receiving cancer treatment (not including carcinoma-in-situ or basal cell cancer of the skin)
* Cirrhosis or end-stage liver disease
* Rheumatologic or chronic inflammatory disease (e.g., systematic lupus erythematous, psoriasis, rheumatoid arthritis, vasculitis, sarcoidosis, Crohn's disease)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Baker, M.D., Principal Investigator — Hennepin Healthcare Research Institute
Locations (4):
- United States (4):
  - UCSF, San Francisco, California
  - NIH Clinical Center, Bethesda, Maryland
  - Allina Health, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota

REFERENCES:
- [Derived] Baker JV, Wolfson J, Collins G, Morse C, Rhame F, Liappis AP, Rizza S, Temesgen Z, Mystakelis H, Deeks S, Neaton J, Schacker T, Sereti I, Tracy RP. Losartan to reduce inflammation and fibrosis endpoints in HIV disease. AIDS. 2021 Mar 15;35(4):575-583. doi: 10.1097/QAD.0000000000002773. PMID 33252490

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Losartan): Participants receive Losartan 100mg daily
- Placebo: Participants receive a matching placebo daily
Period: Overall Study
Arm/Group | Treatment (Losartan) | Placebo
Started | 52 | 56
Completed | 50 | 55
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Losartan) | Placebo | Total
Number analyzed (Participants) | 52 | 56 | 108
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 57 [53 to 62] | 57 [54 to 61] | 57 [54 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 50 | 54 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 4 | 2 | 6
  Not Hispanic - Black | 15 | 22 | 37
  Not Hispanic - White | 31 | 29 | 60
  Not Hispanic - Other | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 52 | 56 | 108
IL-6 [Median (Inter-Quartile Range); unit: pg/mL] | 0.91 [0.67 to 1.3] | 1.04 [.75 to 1.41] | 0.97 [.7 to 1.39]

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin 6 (IL-6) Plasma Levels From Baseline to 12 Months
Description: Difference between treatment and control IL-6 plasma levels from pre-treatment to on-treatment values
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 52 | 56
pg/mL | 0.14 (1.22) | 0.29 (1.25)

2. Secondary Outcome: Change in CD4+ Cell Count From Baseline to 12 Months.
Description: Change in cluster of differentiation 4 (CD4+) cell count from baseline to 12 months
Time Frame: Baseline and 12 months
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | Treatment (Losartan) | Placebo
Number analyzed (Participants) | 52 | 56
Cells/mm^3 | 15.1 (7.6) | 6.8 (7.3)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Treatment (Losartan): Losartan 100mg provided daily
- Placebo: Matching placebo provided daily
Arm/Group | Treatment (Losartan) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/56
Serious Adverse Events (participants affected / at risk) | 6/52 | 4/56
Other Adverse Events (participants affected / at risk) | 22/52 | 13/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Losartan) (N=52) | Placebo (N=56)
Mesenteric Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) — Resolved
Ischaemic Stroke (Vascular disorders) | 0 (0) | 1 (1) — Resolved with sequelae
Hypoglossal Nerve Disorder (Vascular disorders) | 1 (1) | 0 (0) — Chronic, not expected to resolve
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Not resolved
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — Resolved
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Resolved
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Resolved
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Resolved
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Resolved
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Resolved
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Losartan) (N=52) | Placebo (N=56)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 0 (0) | 1 (1)
Ligament Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (3) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Somnambulism (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Gastrointestinal disorders) | 2 (2) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Leukopenia (Immune system disorders) | 1 (1) | 0 (0)
Diabetes Mellitus Type 2 (Endocrine disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT02049307/Prot_SAP_ICF_000.pdf